CLINICAL TRIAL: NCT01886456
Title: Effect of Patterned Laser Trabeculoplasty on Intraocular Pressure Compared to Selective Laser Trabeculoplasty in Treatment Naiv Patients Suffering From Open-angle Glaucoma or Ocular Hypertension
Brief Title: IOP Lowering Effect of PLT Versus SLT in Naiv OAG Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14.1.2013_KEK ZH 2012-0422
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Open Angle Glaucoma,; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

ARMS (2):
- PLT (Experimental): patients treated with patterned laser trabeculoplasty
  Interventions: Device: Laser trabeculoplasty
- SLT (Active Comparator): patients treated with selective laser trabeculoplasty
  Interventions: Device: Laser trabeculoplasty

INTERVENTIONS:
Device: Laser trabeculoplasty

SUMMARY:
To investigate the effect of patterned laser trabeculoplasty (PLT) compared to selective laser trabeculoplasty (SLT) on intraocular pressure (IOP) in treatment naiv patients suffering from open-angle glaucoma or ocular hypertension.

Values for IOP will be measured at baseline, 1 day and 1 month post-interventional as well as 2, 3, 6, 9, 12, 18 and 24 months after treatment.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* Intraocular pressure (treatment naiv or after 4 weeks wash-out phase) > 21 mm Hg
* visible angle structures over 360° on gonioscopy
* age = 18 years

Exclusion criteria:

* Intraocular Inflammation
* patients who underwent refractive corneal surgery for any reason or who underwent ocular surgery to reduce intraocular pressure (e.g. trabeculectomy)
* monocle situation
* anterior chamber lenses (incl. iris claw)
* secondary glaucoma (with the exception of pseudoexfoliation and pigment dispersion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure 6 months after Intervention | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kniestedt, MD, Principal Investigator — University Hospital Zurich, Ophthalmology Clinic
Locations (1):
- University Hospital Zurich, Ophthalmology Clinic, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114